CLINICAL TRIAL: NCT06242821
Title: Back Pain Management in AIS: Impact of Yoga as Adjunct Treatment
Brief Title: Yoga for Back Pain in Adolescent Scoliosis
Acronym: AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00423950
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Scoliosis Idiopathic Adolescent Treatment; Scoliosis Idiopathic; Scoliosis; Adolescence; Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; yoga
MeSH Terms: conditions — Scoliosis | interventions — Standard of Care; Yoga

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate efficacy of a yoga-based intervention as an adjunct treatment for non-operative AIS patients, focusing on those who are braced and non-braced. This clinical trial seeks to provide valuable insights into alternative non-surgical treatment options for AIS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yoga Braced (Active Comparator): Patients, who are currently wearing a brace, are randomized into the yoga group will partake in an online 20 min yoga class 2 days per week
  Interventions: Other: Yoga
- Yoga - Not Braced (Active Comparator): Patients, who are currently not wearing a brace, are randomized into the yoga group will partake in an online 20 min yoga class 2 days per week
  Interventions: Other: Yoga
- Braced - Standard of care (Active Comparator): Patients who are braced, will be randomized into a group that will continue with their standard of care current treatment,
  Interventions: Other: Standard of Care (SOC)
- Non Braced - Standard of care (Active Comparator): Patients who are not braced, will be randomized into a group that will continue with their standard of care current treatment
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Standard of Care (SOC) — Patients will continue with their current standard of care treatment.
  Arms: Braced - Standard of care; Non Braced - Standard of care
Other: Yoga — Patients will be randomized to participate in the Yoga intervention. This will consist of online 20 min yoga classes, 2 times per week. The class will be a set protocol, and patients will be given the protocol to do at home if desired.
  Arms: Yoga - Not Braced; Yoga Braced

SUMMARY:
The Problem: Adolescent Idiopathic Scoliosis (AIS), the pre-eminent spinal pathology affecting over 5% of children and adolescents, presents a pronounced spinal curvature exceeding 10 degrees, with prevalence amongst female adolescents at a ratio of 3:1 compared to males. A significant portion of these patients are not immediate candidates for surgical intervention. The acute shortage of viable non-operative management strategies, which is becoming increasingly imperative given the current barriers to physical therapy access and the growing opioid crisis. The investigator's research intends to explore the addition of a structured yoga protocol to standard of care. This research will thus explore the potential for improved relief and quality-of-life improvements for AIS patients not ready for surgery.

Significance: AIS is a pervasive condition which correlates with chronic and episodic lower back pain, diminished sleep quality, and depressive symptoms. This extensive comorbid association coupled with the financial pressure to patients and the healthcare system cannot be understated.

Needs Statement: There is a lack of sufficient non-operative management options for AIS. Many patients face limited access and require supplementary management strategies to address the patient's conditions effectively, creating a significant unmet need for non-pharmacological pain management interventions. This need is further highlighted in the context of the escalating opioid crisis, a leading cause of death among adolescents and young adults.

Hypothesis: The introduction of a structured yoga protocol can serve as a non-inferior or even superior alternative to traditional standard of care i management of AIS, addressing both the physical and psychosocial aspects intertwined with the condition.

IMPACT: Change in Problem Significance: This research trial aims to enhance current standard of care for patients grappling with AIS. If the trial demonstrates superiority of yoga, it will delineate a paradigm shift in the current care standards for AIS patients, fostering a move towards a more cost-effective and holistic approach. Yoga could help alleviate the burdens on the healthcare system by reducing costs and enhancing accessibility for patients.

Improvement in Pediatric Orthopedics Practice: By paving the way for non-pharmacological interventions, the trial aspires to mitigate the reliance on opioids for pain management in the pediatric demographic, therefore promoting overall well-being. This project not only seeks to develop alternative pain management strategies amidst a growing opioid epidemic but also champions the cause of improving the quality of life for the pediatric population battling chronic conditions like AIS. It echoes the urgent call to innovate and expand upon the current strategies in place, steering the medical community towards a future where integrative approaches are not the exception but the norm. Ultimately, this research aspires to guide the trajectory of pediatric orthopedics towards a healthcare system that is more inclusive, accessible, and holistically oriented, thereby enhancing the quality of life for pediatric patients grappling with conditions like AIS.

2. Objectives (include all primary and secondary objectives) Goals/Objectives: To create a randomized clinical trial aimed to evaluate the efficacy of yoga in conjunction with standard of care treatments for AIS patients.

SPECIFIC AIMS Aim 1: Evaluate the feasibility and challenges of implementing a yoga protocol for AIS patients.

Methodology: Online class attendance, survey completions, and follow-up appointments.

Anticipated Results: Adequate participant adherence and data reliability.

Aim 2: Compare clinical outcomes between patients who receive traditional care modalities versus those who added yoga to treatment plan.

Methodology: Utilize validated tools such as the SRS-22 questionnaire and monitor outcomes including depression scale, sleep quality, analgesic usage, activity levels, and Cobb angle.

Anticipated Results: Significant physical and psychological improvements in the yoga group.

DETAILED DESCRIPTION:
Scoliosis, the most prevalent spinal pathology in children and adolescents, is characterized by a coronal plane spinal curvature more than 10 degrees. Adolescent Idiopathic Scoliosis (AIS) is estimated to impact upwards of 5% of the population with a 3:1 female to male ratio. Treatment options are dictated by curve magnitude and future growth potential. Observation, bracing, supportive physical therapy may be recommended. Research has consistently demonstrated an increasing prevalence of low back pain (LBP) in both children and adolescents over the last few decades. Recent meta-analysis showed that amongst adolescence with LBP, scoliosis is the highest associated abnormality. In addition, biopsychosocial factors are also highly associated with the presence of back pain amongst the AIS population. AIS has been shown to be significantly associated with decreased sleep quality, and depression that is coupled with chronic and/or episodic LBP. This research suggests that patients with AIS should have a psychosocial profile in addition to curve magnitude, and LBP level monitoring.

According to the National Health Interview Survey, 20% of alternative health practitioners state that the practitioners participate in yoga classes for general back pain. The popularity of yoga in the US has increased to an estimated 35 million in 2017, and has become the most utilized complementary health approach. Results of these studies support not only physiological improvement in flexibility, relaxation, and body awareness, but also reduces oxidative stress and inflammation, increases release of neurotransmitters, anxiety and increases pain tolerance resulting in psychological improvement as well. The investigator's study will utilize a well-define a twenty-minute yoga protocol that will be added to some patients undergoing symptomatic non-operative scoliosis treatment. The investigators will measure the angle to see if there is change, the investigator's primary focus will be on reduction of back pain in AIS.

This study consists of a randomized clinical trial with non-operative AIS patients at Johns Hopkins Hospital. The trial will consist of two branches of non-operative AIS patients: 1. Patients that brace, 2. Patients who do not brace. This allocation will be achieved through random assignment to either the patient's standard of care as prescribed with or without the addition of yoga.

ELIGIBILITY:
Inclusion Criteria:

* Non-operatively treated AIS patients at Johns Hopkins Hospital with back pain who are candidates for physical therapy.
* Cobb angle: greater than 25 degrees,
* Visual Analog Scale (VAS) Pain score greater than 41/0
* Braced and Unbraced Patients

Exclusion Criteria:

* Scoliosis due to causes other than AIS.
* AIS patients who have undergone surgery for scoliosis or back pain
* Age less than 10 years of age or greater than 20 years of age
* Unable to access zoom on any electronic device

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain and Quality of Life as assessed by the Scoliosis Research Society (SRS-22) questionnaire | Enrollment, 6 months, 1 year
  Possible score range from 0 (no pain)to 5(worst possible pain). A higher score indicates a better quality of life.
Participant Engagement | Enrollment, 6 months, 1 year
  Participant engagement will be measured by comparing attendance and adherence rates between the two groups to assess patient engagement with each intervention.

SECONDARY OUTCOMES:
Cobb Angle measurement | Enrollment, 6 months, 1 yr
  Patients will have cobb angle (extent of scoliotic curve) measured

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sponseller, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No